CLINICAL TRIAL: NCT02105415
Title: Ketamine / Propofol Admixture "Ketofol" at Induction in the Critically Ill Against Etomidate: KEEP PACE Trial
Acronym: KEEP PACE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nathan J. Smischney, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-000506
Record Dates: First submitted 2014-03-31; First posted 2014-04-07 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Critical Illness
Keywords: Critical care; Emergent; Etomidate; Hemodynamics; Intensive care unit; Intubation; Ketamine-Propofol admixture
MeSH Terms: conditions — Critical Illness | interventions — Ketamine; Etomidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etomidate (Active Comparator): weight based dose of 0.15mg/kg
  Interventions: Drug: Etomidate
- Ketamine / Propofol Admixture (Experimental): weight based dose of 0.5mg/kg of ketamine and 0.5mg/kg of propofol
  Interventions: Drug: Ketamine / Propofol Admixture

INTERVENTIONS:
Drug: Ketamine / Propofol Admixture
  Arms: Ketamine / Propofol Admixture
Drug: Etomidate
  Arms: Etomidate

SUMMARY:
The hypothesis of this study is that a Ketamine / Propofol mixture will produce more stable hemodynamics as compared to Etomidate during emergent intubations in the intensive care unit. Patients that require a breathing tube to be placed in the ICU will be randomized to receIve either a Ketamine / Propofol mixture or Etomidate for sedation in order to place the breathing tube.

DETAILED DESCRIPTION:
Endotracheal intubation is a procedure that may cause significant hemodynamic perturbations and can severely impact the outcome of the critically ill. To ensure a safe outcome during this particular procedure, there are many factors that the clinician is faced with. One decision that confronts the critical care physician involves the correct combination of medications with which to facilitate such a safe outcome. Given the reported hemodynamic stability, etomidate is a medication that is chosen by many providers in this particular situation. However, its association with a possible increase in mortality makes it less than ideal for a number of critical care physicians. In recent years, an admixture of propofol and ketamine has been studied that demonstrates hemodynamic stability based on the balancing of the hemodynamic effects of these two individual agents alone. This novel medication combination, sometimes referred to as "ketofol", may offer a valuable alternative to the critical care physician. Therefore, a randomized parallel-group clinical trial of adult critically ill patients admitted to a medical and/or surgical intensive care unit at Mayo Clinic Rochester who meet the criteria designated below for which urgent and/or emergent intubation is needed will receive one of two interventions based on stratified randomization. The "active" intervention arm will receive ketamine/propofol (ketofol) to facilitate endotracheal intubation. The comparison arm will receive etomidate. The primary outcome will focus on hemodynamic data recorded during the first 5 minutes post-administration with secondary outcomes looking at hemodynamic data at 10 and 15 minutes and addressing intensive care unit length of stay, mortality, adrenal function, and vasoactive medication use, among others.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Surgical or medical intensive care unity patients requiring endotracheal intubation
* Consulting physician agrees to study plan and will follow drug randomization

Exclusion Criteria:

* Known intracranial pathology
* Known chronic opiate-dependence
* Received continuous sedative infusion in the last 24 hours
* Known severe psychiatric illness
* Known egg allergies
* Known contraindication to fentanyl, midazolam, ketamine, propofol or etomidate
* Intubation in which standard practice is not to use sedation
* No known documented weight or weight greater than 140 kg or less than 30 kg
* Prior participation in the study
* Of childbearing age (18-50) with no known negative pregnancy test on this admission.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-04; Primary Completion 2017-11-28 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Smischney, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Smischney NJ, Seisa MO, Schroeder DR. Association of Shock Indices with Peri-Intubation Hypotension and Other Outcomes: A Sub-Study of the KEEP PACE Trial. J Intensive Care Med. 2024 Sep;39(9):866-874. doi: 10.1177/08850666241235591. Epub 2024 Feb 25. PMID 38403984
- [Derived] Smischney NJ, Nicholson WT, Brown DR, Gallo De Moraes A, Hoskote SS, Pickering B, Oeckler RA, Iyer VN, Gajic O, Schroeder DR, Bauer PR. Ketamine/propofol admixture vs etomidate for intubation in the critically ill: KEEP PACE Randomized clinical trial. J Trauma Acute Care Surg. 2019 Oct;87(4):883-891. doi: 10.1097/TA.0000000000002448. PMID 31335755
- [Derived] Smischney NJ, Hoskote SS, Gallo de Moraes A, Racedo Africano CJ, Carrera PM, Tedja R, Pannu JK, Hassebroek EC, Reddy DR, Hinds RF, Thakur L. Ketamine/propofol admixture (ketofol) at induction in the critically ill against etomidate (KEEP PACE trial): study protocol for a randomized controlled trial. Trials. 2015 Apr 21;16:177. doi: 10.1186/s13063-015-0687-0. PMID 25909406

RESULTS

PARTICIPANT FLOW:
Groups:
- Etomidate: Etomidate 0.15mg/kg weight based dose
- Ketamine / Propofol Admixture: Ketamine / Propofol Admixture; weight based dose 0.5 mg/kg ketamine and 0.5 mg/kg propofol.
Period: Overall Study
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Started | 76 | 84
Completed | 73 | 79
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Ketamine / Propofol Admixture: Ketamine / Propofol Admixture weight based dose 0.5 mg/kg ketamine and 0.5 mg/kg propofol
- Total: Total of all reporting groups
Arm/Group | Etomidate | Ketamine / Propofol Admixture | Total
Number analyzed (Participants) | 73 | 79 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (18.3) | 62.1 (17.2) | 61.1 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 38 | 48 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 57 | 76 | 133
  Unknown or Not Reported | 16 | 3 | 19
Region of Enrollment [Number; unit: participants]
  United States | 73 | 79 | 152

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure
Description: Mean arterial pressure for the ketamine/propofol group at a 1:1 dose ratio compared to the etomidate group within the first 15 minutes post-administration in patients in need of urgent and/or emergent endotracheal intubation, as defined by any intubation within the intensive care unit excluding intubations for elective procedural events and codes.
Time Frame: baseline and every 5 minutes up to 15 minutes minutes post study drug administration
Population: Data are presented for patients who had blood pressure measurements at baseline (within 15 minutes prior to study drug administration).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Number analyzed (Participants) | 70 | 76
mm Hg
  Baseline | 82.8 (17.9) | 80.9 (13.3)
  5 minutes: number analyzed (Participants) | 69 | 75
  5 minutes | 81.7 (17.2) | 77.6 (15.4)
  10 minutes: number analyzed (Participants) | 67 | 69
  10 minutes | 81.9 (20.0) | 75.3 (20.3)
  15 minutes: number analyzed (Participants) | 68 | 70
  15 minutes | 79.1 (19.5) | 75.5 (18.1)
Statistical Analysis 1: Comparison: Etomidate vs Ketamine / Propofol Admixture; 5 minutes; Test type: Superiority; p = 0.385, ANCOVA; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-6.9 to 2.7]
Statistical Analysis 2: Comparison: Etomidate vs Ketamine / Propofol Admixture; 10 minutes; Test type: Superiority; p = 0.241, ANCOVA; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-10.8 to 2.8]
Statistical Analysis 3: Comparison: Etomidate vs Ketamine / Propofol Admixture; 15 minutes; Test type: Superiority; p = 0.802, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-7.2 to 5.6]

2. Secondary Outcome: Mortality
Description: In-hospital/28 day mortality among patients in ketamine/propofol combination compared to in-hospital/28-day mortality in etomidate.
Time Frame: Hospital Discharge or Day 28, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Number analyzed (Participants) | 73 | 79
Participants | 26 | 25
Statistical Analysis 1: Comparison: Etomidate vs Ketamine / Propofol Admixture; Test type: Superiority; p = 0.605, ANCOVA

3. Secondary Outcome: Vasopressor Use
Description: The use of vasoactive medications to restore the blood pressure post-administration in the ketamine/propofol combination as compared to the etomidate group.
Time Frame: up to 24 hours post study drug administration
Population: Data are presented for patients who had vasopressor data within the time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Number analyzed (Participants) | 73 | 79
Participants
  Pre-treament | 1 | 5
  New-onset pressors (within 3 minutes): number analyzed (Participants) | 72 | 76
  New-onset pressors (within 3 minutes) | 12 | 18
  Delayed-onset pressors (within 24 hours) | 57 | 64
Statistical Analysis 1: Comparison: Etomidate vs Ketamine / Propofol Admixture; Pre-treatment; Test type: Superiority; p = 0.212, ANCOVA
Statistical Analysis 2: Comparison: Etomidate vs Ketamine / Propofol Admixture; New-onset pressors (within 3 minutes); Test type: Superiority; p = 0.308, ANCOVA
Statistical Analysis 3: Comparison: Etomidate vs Ketamine / Propofol Admixture; Delayed-onset pressors (within 24 hrs); Test type: Superiority; p = 0.691, ANCOVA

4. Secondary Outcome: Number of Participants With Adrenal Insufficiency
Description: Incidence of adrenal insufficiency between ketamine/propofol admixture and etomidate. Adrenal insuffiency was evaluated with co-syntropin stimulation test.
Time Frame: up to 24 hours post study drug administration
Population: A secondary outcome included adrenal testing in a subset of patients. Thus, cortisol levels were available for 29 subjects at 3 and 5 hours and 30 subjects at 23 and 25 hours.
Measure: Count of Participants; unit: Participants
Groups:
- Etomidate (3-5 Hours); Ketamine/Propofol Admixture (3-5 Hours): Cortisol levels at 3-5 hours
- Etomidate (23-25 Hours); Ketamine/Propofol Admixture (23-25 Hours): Cortisol levels at 23-25 hours
Arm/Group | Etomidate (3-5 Hours) | Ketamine/Propofol Admixture (3-5 Hours) | Etomidate (23-25 Hours) | Ketamine/Propofol Admixture (23-25 Hours)
Number analyzed (Participants) | 16 | 13 | 15 | 15
Participants | 13 | 5 | 9 | 6

5. Secondary Outcome: Mechanical Ventilation Free Days
Description: comparison of mechanical ventilation free days between the two groups
Time Frame: hospital discharge or day 28, whichever comes first
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Number analyzed (Participants) | 73 | 79
days | 22 [0 to 25] | 20 [0 to 26]
Statistical Analysis 1: Comparison: Etomidate vs Ketamine / Propofol Admixture; Test type: Superiority; p = 0.911, ANCOVA

6. Secondary Outcome: Blood Product Transfusions
Description: blood product transfusions [Red Blood Cells vs. non-Red Blood Cells] between the two groups
Time Frame: hospital discharge or day 28, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Number analyzed (Participants) | 73 | 79
Participants
  Red blood cell | 21 | 13
  Non-red blood cell | 16 | 8
  Colloid | 28 | 26
Statistical Analysis 1: Comparison: Etomidate vs Ketamine / Propofol Admixture; Red blood cell; Test type: Superiority; p = 0.069, ANCOVA
Statistical Analysis 2: Comparison: Etomidate vs Ketamine / Propofol Admixture; Non-red blood cell; Test type: Superiority; p = 0.046, ANCOVA
Statistical Analysis 3: Comparison: Etomidate vs Ketamine / Propofol Admixture; Colloid; Test type: Superiority; p = 0.502, ANCOVA

7. Secondary Outcome: Intensive Care Unit Free Days
Description: comparison of intensive care unit free days between the two groups
Time Frame: hospital discharge or day 28, whichever comes first
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Number analyzed (Participants) | 73 | 79
days | 16 [0 to 23] | 17 [0 to 24]
Statistical Analysis 1: Comparison: Etomidate vs Ketamine / Propofol Admixture; Test type: Superiority; p = 0.994, ANCOVA

8. Secondary Outcome: Number of Participants Experiencing Delirium Using Confusion Assessment Method in ICU
Description: Comparison of number of participants who were positive for delirium using CAM-ICU between groups
Time Frame: up to 24 hours post study drug administration
Population: The analysis of new onset delirium was restricted to subjects (54 etomidate, 62 KPA) who did not experience delirium pre-study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine / Propofol Admixture
Number analyzed (Participants) | 54 | 62
Participants | 7 | 4
Statistical Analysis 1: Comparison: Etomidate vs Ketamine / Propofol Admixture; Test type: Superiority; p = 0.233, ANCOVA

ADVERSE EVENTS:
Time Frame: Given the context of the study and the emergent nature in which the interventions were conducted, adverse events were collected up to 72 hours after enrollment.
Arm/Group | Etomidate | Ketamine / Propofol Admixture
All-Cause Mortality (participants affected / at risk) | 26/73 | 25/79
Serious Adverse Events (participants affected / at risk) | 6/73 | 5/79
Other Adverse Events (participants affected / at risk) | 19/73 | 14/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etomidate (N=73) | Ketamine / Propofol Admixture (N=79)
Cardiac arrest (Cardiac disorders) | 0 | 2
Hypertensive urgency (Vascular disorders) | 2 | 0
Severe hypotension (Vascular disorders) | 4 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etomidate (N=73) | Ketamine / Propofol Admixture (N=79)
Intubation Complication (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
IV infiltration (General disorders) | 2 (2) | 0 (0)
Multi organ failure (General disorders) | 4 (4) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vomiting/Aspiration (General disorders) | 3 (3) | 2 (2)
arrythmia (Cardiac disorders) | 1 (1) | 0 (0)
shock (Vascular disorders) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
Single center study with non-blinded interventions and non-controlled co-interventions all of which can impact hemodynamics. Selection bias with 92 non-enrollees.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT02105415/Prot_SAP_000.pdf